CLINICAL TRIAL: NCT02458144
Title: Comparison of Two Minimally Invasive Approaches to the Hip-anterior Versus Anterolateral - Which Technique is Less Invasive? A Prospective, Randomized, Controlled Pilot Study
Brief Title: Comparison of MIS Anterior Versus MIS Anterolateral Approach
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Christoph Stihsen, Dr. med. univ., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1392/2012
Record Dates: First submitted 2015-05-26; First posted 2015-05-29 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Osteoarthritis of the Hip
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MIS "anterior" group (Other): Total Hip Arthroplasty "anterior" surgical approach
  Interventions: Procedure: Total hip arthroplasty
- MIS "anterolateral" group (Other): Total Hip Arthroplasty "anterolateral" surgical approach
  Interventions: Procedure: Total hip arthroplasty

INTERVENTIONS:
Procedure: Total hip arthroplasty — The minimally invasive anterior approach The patient is in supine position. The femoral neck is exposed in the interval between tensor fasciae latae, glutei medius and minimus muscles laterally, and sartorius and rectus femoris muscles medially. After osteotomy of the neck and extraction of the head the acetabulum is reamed to prepare for cup prosthesis. Following peritrochanteric capsulotomy the externally rotated, adducted and elevated femur is broached.
  The MIS anterolateral approach The MIS anterolateral technique is a modified Watson-Jones Approach. The patient is in supine position. This approach uses the intermuscular plane between the gluteus medius and the tensor fascia latae. After the anterior capsule is excised, a disc of the femoral neck is removed.

SUMMARY:
Aim of the present investigation is to analyse the amount of muscle trauma in relation to the surgical approach and to the individual postoperative functional recovery. The investigation will compare the MIS (minimally invasive surgery) anterior approach with the MIS anterolateral approach to the hip.

DETAILED DESCRIPTION:
The surgical approach to the hip is reportedly an important factor influencing implant stability and postsurgical muscle functioning. Reviewing the literature, controversial studies towards minimally invasive hip surgery can be found. Currently, none of the approaches can be considered superior, but the trend is towards minimally invasive techniques, as it is generally accepted that muscle trauma and damage of the periarticular structures should be minimized. However, a surgical approach that causes no damage to surrounding muscle is unrealistic. Whether the muscle is stretched, transacted or partially torn, injury will occur.

Aim of the present investigation is to analyse the amount of muscle trauma in relation to the surgical approach and to the individual postoperative functional recovery. The investigation will compare the MIS anterior approach with the MIS anterolateral approach to the hip. The investigators questioned, which technique would be the less invasive? Pain and functional performance will be measured using the Harris Hip Score, the Western Ontario McMaster, and the UCLA (University of California) Activity Score. Subject quality-of-life will be determined by evaluation the Short-Form 36 Health Survey. Standard radiographs of the hip are required to be captured before surgery and at 3, 6 and 12 months postoperatively. MRI scans will be performed to evaluate tendon defects, fatty atrophy and changes in the muscle cross-sectional area. Next, the patients will be referred for hip sonography, performed by a radiologist who is experienced in imaging of the musculoskeletal system who will be unaware of the clinical examination results of the patients. Moreover gait analyses will be performed preoperatively, 3 and 12 months after surgery. Pre- and postoperative standard blood tests and specific serum trauma markers will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* unilateral, noninflammatory end-stage osteoarthritis of the hip
* willingness and ability to cooperate in the required post-operative therapy
* willingness and ability to provide written informed consent
* age 50-80 years

Exclusion Criteria:

* inflammatory arthropathies
* prior hip surgery
* prior infection of the hip
* severe morbidity
* severe osteoporosis
* inability to tolerate general anesthesia
* no contraindications to MRI e.g. pacemakers, claustrophobia
* neuromuscular disorder, vascular disorder or other conditions that could contribute to prosthesis instability, prosthesis fixation failure, or complications in postoperative care
* known alcohol or drug abuse
* unwillingness to participate

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-08 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
MRI evaluation | 12 months after surgery
  Cross-sectional area of gluteus medius and tensor fascia latae muscle (cm2)

SECONDARY OUTCOMES:
Harris Hip Score | 12 months after surgery
  Points (0-100)
Tendon defects of the hip abductors (cm) assessed by Ultrasound | 12 months after surgery
  Tendon defects of the hip abductors (cm)
Gait analysis | 12 months after surgery
  posture of the pelvis, hip strength, range of motion
Serum trauma marker 1 | 1 hour preop. to 48 hours postop.
  creatinkinase (u/l)
Serum trauma marker 2 | 1 hour preop. to 48 hours postop.
  interleukin-6 (pg/ml)
Serum trauma marker 3 | 1 hour preop. to 48 hours postop.
  interleukin-1β (pg/ml)
Serum trauma marker 4 | 1 hour preop. to 48 hours postop.
  lactate Dehydrogenase (u/l)
Serum trauma marker 5 | 1 hour preop. to 48 hours postop.
  aldolase (u/l)
Serum trauma marker 6 | 1 hour preop. to 48 hours postop.
  Myoglobin (ng/ml)
Serum trauma marker 7 | 1 hour preop. to 48 hours postop.
  malondialdehyde (mg/dl)
Serum trauma marker 8 | 1 hour preop. to 48 hours postop.
  glutathione (mg/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Reinhard Windhager, Chairman, Study Chair — Medical University of Vienna
Locations (1):
- Department of Orthopaedics, Vienna, Vienna, Austria